CLINICAL TRIAL: NCT01065740
Title: Optimized Supervised Education Program for Peripheral Arterial Disease: Ambulatory Management With Patient Education
Brief Title: Optimized Supervised Education Program for Peripheral Arterial Disease
Acronym: POPART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Difficulties and Financing Limited and exhausted
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: phrq/09-01
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Patient education; Physical activity coaching; Lifestyle modifications; Walking capacity; 6 minutes walking test
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient education (Experimental): individual and group meetings with explanations about the disease, lifestyle counseling ; coaching by phone at 1 and 4 months; medical consultation at 3 months; physical exercise with coaching
  Interventions: Other: Patient education
- Usual care (No Intervention)

INTERVENTIONS:
Other: Patient education
  Arms: patient education

SUMMARY:
Peripheral arterial disease (PAD) is a frequent and serious chronic disease witch is undertreated. The recommended management of PAD include pharmacological approach and lifestyle modifications. Patient education help to reach this outcome. Our study propose to compare patient education management with physical activity coaching to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years
* With peripheral arterial disease
* Who accept to follow a patient education program

Exclusion Criteria:

* Permanent limb ischemia
* Revascularisation programmed in the 6 next months
* Other severe prognostic disease
* Difficulties to obtain patient consent because of language or understanding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
6 minutes walking test | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France